CLINICAL TRIAL: NCT00207740
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study Evaluating the Efficacy and Safety of CNTO 148 Administered Subcutaneously in Symptomatic Subjects With Severe Persistent Asthma
Brief Title: A Study of Safety and Efficacy of CNTO 148 in Patients With Severe Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Centocor BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005281; C0524T03 (Other: Centocor)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
Keywords: Asthma; Severe Persistent Asthma; Subcutaneous injections; Immunology disorder; Breathlesness
MeSH Terms: conditions — Asthma | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CNTO 148 (golimumab) (Experimental)
  Interventions: Drug: CNTO148
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNTO148 — Type=exact type, unit=mg, number=50, 75, 100, 150, 200 and 300, form=injection, route=subcutaneous. Every 4 weeks partciapnts will receive injections in 4 parallel treatment arms
  Arms: CNTO 148 (golimumab)
Drug: Placebo — Type=exact type, unit=mg, form=injection, route=subcutaneous. Placebo will be given from from Week 0 through Week 52.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of CNTO 148 (golimumab) in patients with severe persistent asthma.

DETAILED DESCRIPTION:
This is a multicenter, randomized (the study medication is assigned by chance), double-blind (neither physician nor patient knows the treatment that the patient receives), placebo-controlled (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical study), parallel-group (each group of patients will be treated at the same time), dose-ranging study to evaluate the efficacy and safety of CNTO 148. The study will consists of run-in phase (2 weeks), treatment period (52 weeks) and follow up period (24 weeks). The patients inhaled corticosteroids (ICS) medication will be standardized in the run-in phase and the treatment period contains first 24 weeks of treatment, the patients are required to remain on stable doses of concomitant corticosteroids (CS) medication (steroid stable phase). The steroid stable phase is followed by a 28-week steroid taper phase, during which a reduction of concomitant CS medication will be attempted. After completion of the study treatment, patients are to be followed for an additional 24 weeks. Patients will receive subcutaneous injections of 75, 150, or 300 mg of CNTO 148 or placebo every 4 weeks for 52 weeks followed 50,100, or 200 mg every 4 weeks through week 52. The safety of the patient will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma for greater than or equal to 3 years and a diagnosis of severe persistent asthma forgreater than or equal to 1 year prior to screening
* Continuous treatment with high dose Inhaled corticosteroids (ICS) and long acting beta-agonist for at least 3 months prior to screening
* Have evidence of at least 1 of the following in the 5 years prior to screening or during screening, reversible airway obstruction greater than or equal to 12 percentage change in forced expiratory volume in 1 second (FEV1) postbronchodilator; Diurnal variation in peak expiratory flow rate (PEFR) greater than or equal to 30 percentage change) and airway hyperresponsiveness
* Estimated frequency of symptoms on more than one-third of days for at least 3 months prior to screening (eg, wheezing, breathlessness, chest tightness, cough, nocturnal awakening) despite treatment with high dose ICS and long-acting β2-agonist (LABA), with or without continuous oral corticosteroids
* Score of greater than or equal to 2 points on the asthma control questionnaire at screening.

Exclusion Criteria:

* Diagnosis of chronic obstructive pulmoanry disease (COPD), cystic fibrosis, or other significant respiratory disorder
* Worsening of asthma symptoms that required treatment with an addition or increase in oral corticosteroids dose (steroid burst) in the 4-week period prior to the screening visit
* Life-threatening asthma attack requiring cardiopulmonary support (eg, intubation) in the 6-month period prior to screening
* Have ever used alkylating agents (eg, chlorambucil or cyclophosphamide)
* Concomitant diagnosis or any history of congestive heart failure (CHF), including medically controlled CHF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2004-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (57):
- United States (29):
  - Los Angeles, California
  - San Diego, California
  - Stockton, California
  - Denver, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Chicago, Illinois
  - Normal, Illinois
  - River Forest, Illinois
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - North Dartmouth, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Cortland, New York
  - Elmira, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Lake Oswego, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - El Paso, Texas
  - Richmond, Virginia
  - Bellingham, Washington
  - Madison, Wisconsin
- Ghent, Belgium
- Bulgaria (2):
  - Russel
  - Sofia
- Czechia (3):
  - Ostrava
  - Poruba
  - Ústí nad Labem
- France (3):
  - Montpellier
  - Pessac
  - Tarbes
- Germany (4):
  - Berlin
  - Großhansdorf
  - Leipzig
  - Mainz
- Hungary (5):
  - Budapest
  - Nyíregyháza
  - Székesfehérvár
  - Szombathely
  - Törökbálint
- Leiden, Netherlands
- Poland (5):
  - Bieńkówka
  - Katowice
  - Lodz
  - Torun
  - Warsaw
- Sweden (2):
  - Linköping
  - Stockholm
- United Kingdom (2):
  - Glasgow
  - Southampton

REFERENCES:
- [Derived] Wenzel SE, Barnes PJ, Bleecker ER, Bousquet J, Busse W, Dahlen SE, Holgate ST, Meyers DA, Rabe KF, Antczak A, Baker J, Horvath I, Mark Z, Bernstein D, Kerwin E, Schlenker-Herceg R, Lo KH, Watt R, Barnathan ES, Chanez P; T03 Asthma Investigators. A randomized, double-blind, placebo-controlled study of tumor necrosis factor-alpha blockade in severe persistent asthma. Am J Respir Crit Care Med. 2009 Apr 1;179(7):549-58. doi: 10.1164/rccm.200809-1512OC. Epub 2009 Jan 8. PMID 19136369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 309 patients were randomized into 4 parallel treatment groups at 53 sites (134 patients at 27 sites in the US and 175 patients at 26 sites in Europe). The first patient was consented on 31 Aug 2004, and the last patient completed the study on 17 Jul 2007.
Groups:
- Group I: Placebo: Placebo subcutaneous (SC) injections every 4 weeks (Wks) from week (Wk) 0 to Wk 52
- Group II: Golimumab 50 mg: Golimumab (CNTO148) 75 mg SC injection at Wk 0 followed by 50 mg SC injections every 4 Wks to Wk 52
- Group III: Golimumab 100 mg: Golimumab 150 mg SC injection at Wk 0 followed by 100 mg SC injections every 4 Wks to Wk 52
- Group IV: Golimumab 200 mg: Golimumab 300 mg SC injection at Wk 0 followed by 200 mg SC injections every 4 Wks to Wk 52
Period: Overall Study
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg
Started | 78 | 77 | 76 | 78
Completed | 49 (Indicates number of patients who received subcutaneous study medication through Week 52) | 36 (Indicates number of patients who received subcutaneous study medication through Week 52) | 36 (Indicates number of patients who received subcutaneous study medication through Week 52) | 35 (Indicates number of patients who received subcutaneous study medication through Week 52)
Not Completed | 29 | 41 | 40 | 43
Not completed — Adverse Event | 4 | 14 | 14 | 11
Not completed — Unsatisfactory therapeutic effect | 1 | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 2 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Sponsor Directive | 22 | 15 | 16 | 21
Not completed — Other | 2 | 10 | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg | Total
Number analyzed (Participants) | 78 | 77 | 76 | 78 | 309
Age Continuous [Mean (Standard Deviation); unit: years] | 49.4 (12.03) | 49.4 (11.26) | 49.1 (12.85) | 52.7 (12.26) | 50.1 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 46 | 39 | 46 | 173
  Male | 36 | 31 | 37 | 32 | 136

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Prebronchodilator Clinic-Measured, Percent-Predicted Forced Expiratory Volume in 1 Second
Description: The endpoint is change from baseline in prebronchodilator clinic-measured percent predicted Percent-Predicted Forced Expiratory Volume in 1 Second (FEV1) with Last Observation Carried Forward (LOCF) at 6 months. The baseline visit starts at the end of 2 weeks run in phase.
Time Frame: Baseline and Week 24
Population: The analysis of this endpoint uses intent-to-treat population. Missing data were imputed using Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent predicted
Groups:
- Group II: Golimumab 50 mg: Golimumab (CNTO148) 75 milligram (mg) SC injection at Wk 0 followed by 50 mg SC injections every 4 Wks to Wk 52
- Combined: Group III & IV: Combines Group III (golimumab 100 mg) and Group IV (golimumab 200 mg)
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg | Combined: Group III & IV
Number analyzed (Participants) | 78 | 77 | 76 | 78 | 154
Percent predicted | 2.44 [-0.574 to 5.461] | 0.48 [-2.563 to 3.519] | 3.22 [0.149 to 6.295] | 2.59 [-0.441 to 5.620] | 2.91 [0.696 to 5.116]
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group III & IV; The null hypothesis was that the endpoint for placebo is the same as that for combined 100 mg and 200 mg golimumab. Assuming a standard deviation of 23%, there is 86% power to detect a 10% difference at a 0.05 significance level; Test type: Superiority or Other; p = 0.802, ANCOVA — When interpreting this p-value along with the other co-primary endpoint, Hochberg procedure was used
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Golimumab 200 mg; This is a secondary analysis; Test type: Superiority or Other; p = 0.945, ANCOVA — The nominal p-value is for descriptive purpose only
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; This is a secondary analysis; Test type: Superiority or Other; p = 0.717, ANCOVA — The nominal p-value is for descriptive purpose only
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; This is a secondary analysis; Test type: Superiority or Other; p = 0.357, ANCOVA — The nominal p-value is for descriptive purpose only

2. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire Score at 6 Months; Randomized Patients
Description: The endpoint is the change from baseline in the overall Asthma Quality of Life Questionnaire (AQLQ) score at 6 months. The AQLQ is a validated and self-administered questionnaire to evaluate symptoms and Quality of Life (QOL) in subjects with asthma and it has 32 questions in 4 domains (symptoms, activity limitations, emotional function, and environmental stimuli). Participants were asked to score the importance of each of the positively identified problems on a 7-point scale (7 = not impaired at all - 1 = severely impaired).
Time Frame: Baseline to Week 24
Population: The analysis of this endpoint uses intent-to-treat population. Missing data were imputed using last observation carried forward.
Measure: Median (Inter-Quartile Range); unit: Points on scale
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg | Combined: Group III & IV
Number analyzed (Participants) | 78 | 77 | 76 | 78 | 154
Points on scale | 0.42 [0.00 to 1.13] | 0.53 [0.00 to 1.13] | 0.86 [-0.02 to 1.47] | 0.55 [0.00 to 1.00] | 0.66 [0.00 to 1.34]
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group III & IV; The null hypothesis was that the endpoint for placebo is the same as that in the combined 100 mg and 200 mg golimumab; Test type: Superiority or Other; p = 0.286, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Golimumab 200 mg; Test type: Superiority or Other; p = 0.742, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p = 0.128, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p = 0.946, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Number of Severe Asthma Exacerbations Per Patient From Baseline Through 6 Months
Description: The endpoint is the average number of severe asthma exacerbations per patient from baseline through 6 months.
Time Frame: Baseline to Week 24
Population: The analysis of this endpoint uses intent-to-treat population. For the dropouts, the worst case in similar patients was used as the number of severe exacerbations.
Measure: Mean (Standard Deviation); unit: Events per patient through week (Wk) 24
Groups:
- Group II: Golimumab 50 mg: Golimumab 75 milligram (mg) SC injection at Wk 0 followed by 50 mg SC injections every 4 Wks to Wk 52
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg | Combined: Group III & IV
Number analyzed (Participants) | 78 | 77 | 76 | 78 | 154
Events per patient through week (Wk) 24 | 0.5 (1.07) [0.0 to 1.0] | 0.7 (1.18) [0.0 to 1.0] | 0.4 (0.85) [0.0 to 0.5] | 0.5 (1.08) [0.0 to 1.0] | 0.5 (0.97) [0.0 to 1.0]
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group III & IV; The null hypothesis was that the number of severe exacerbations per patient from baseline through week 24 for placebo is the same as that in the combined 100 mg and 200 mg golimumab. Assuming 1 severe exacerbation over 6 months per patient in the placebo group, there is 79% power to detect a 35% reduction in the combined 100 mg and 200 mg golimumab group at a 0.05 significance level; Test type: Superiority or Other; p = 0.718, Cochran-Mantel-Haenszel — When interpreting this p-value along with the other co-primary endpoint, Hochberg procedure was used
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Golimumab 200 mg; This is a secondary analysis; Test type: Superiority or Other; p = 0.779, Cochran-Mantel-Haenszel — The nominal p-value is for descriptive purpose only
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; This is a secondary analysis; Test type: Superiority or Other; p = 0.649, Cochran-Mantel-Haenszel — The nominal p-value is for descriptive purpose only
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; This is a secondary analysis; Test type: Superiority or Other; p = 0.256, Cochran-Mantel-Haenszel — The nominal p-value is for descriptive purpose only

4. Secondary Outcome: Change From Baseline in Rescue Medication Use at 6 Months; Randomized Patients
Description: The endpoint is change from baseline in rescue medication use at Wk 24 where the rescue medication use was based on the average over 7 days prior to visit.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Puffs/day
Groups:
- Group II: Golimumab 50 mg: Golimumab 75 mg SC injection at Wk 0 followed by 50 mg SC injections every 4 Wks to Wk 52
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg | Combined: Group III & IV
Number analyzed (Participants) | 78 | 77 | 76 | 78 | 154
Puffs/day | -0.54 [-1.57 to 0.50] | -0.71 [-1.71 to 0.52] | -0.29 [-1.79 to 0.26] | -0.14 [-1.67 to 0.67] | -0.21 [-1.71 to 0.57]
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group III & IV; The null hypothesis was that the endpoint for placebo is the same as that in the combined 100 mg and 200 mg golimumab; Test type: Superiority or Other; p = 0.894, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Golimumab 200 mg; Test type: Superiority or Other; p = 0.572, Kruskal-Wallis
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p = 0.731, Kruskal-Wallis
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p = 0.856, Kruskal-Wallis

5. Secondary Outcome: Number of Severe Asthma Exacerbations Per Patient From Week 24 Through Week 52; Randomized Patients Who Did Not Discontinue Study Participation Prior to Week 24
Description: The endpoint is the average number of severe asthma exacerbations per patient from Week (Wk) 24 through Wk 52 for the patients who did not discontinue study participation prior to Wk 24
Time Frame: Week 24 to Week 52
Population: Analysis of this endpoint only includes patients (pts) who did not discontinue study participation prior to Wk 24. For the dropouts during the period between Wks 24- 52, worst case in similar pts was used as the number of severe exacerbations. Data from Wk 24-52 must be interpreted with caution as study agent was stopped at various study timepoints
Measure: Mean (Standard Deviation); unit: Events per patient from Wk 24 thru Wk 52
Groups:
- Group I: Placebo: Placebo subcutaneous (SC) injections every 4 weeks (Wks) from Wk 0 to Wk 52
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg | Combined: Group III & IV
Number analyzed (Participants) | 77 | 68 | 71 | 74 | 145
Events per patient from Wk 24 thru Wk 52 | 0.6 (1.02) [0.0 to 1.0] | 0.8 (1.23) [0.0 to 2.0] | 0.9 (1.18) [0.0 to 2.0] | 0.8 (1.01) [0.0 to 2.0] | 0.9 (1.09) [0.0 to 2.0]
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group III & IV; The null hypothesis was that the endpoint for placebo is the same as that in the combined 100 mg and 200 mg golimumab; Test type: Superiority or Other; p = 0.273, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Golimumab 200 mg; Test type: Superiority or Other; p = 0.382, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p = 0.350, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p = 0.341, Cochran-Mantel-Haenszel

6. Secondary Outcome: Change From Baseline in Oral Corticosteroids Dose at Week 52; Randomized Patients Who Received Oral Corticosteroids at Baseline
Description: The endpoint is the change from baseline at Week (Wk) 52 in oral corticosteroids (OCS) dose for the randomized patients who received OCS at baseline.
Time Frame: Baseline and Week 52
Population: Analysis of this endpoint includes only pts who received OCS at baseline.Wk 52 OCS dose is the daily OCS dose in the last period, defined as between 2 consecutive visits, in which no change in total daily dose of OCS occurred, prior to Wk 52 visit.Data from Wk 24-52 must be interpreted with caution as study agent was stopped at various timepoints.
Measure: Median (Inter-Quartile Range); unit: mg/day P. Eq.
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg | Combined: Group III & IV
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 49
mg/day P. Eq. | -5.000 [-10.000 to 0.000] | 0.000 [-5.000 to 0.000] | -4.550 [-10.000 to 0.000] | -3.750 [-10.000 to 0.000] | -4.550 [-10.000 to 0.000]
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group III & IV; The null hypothesis was that the endpoint for placebo is the same as that in the combined 100 mg and 200 mg golimumab; Test type: Superiority or Other; p = 0.986, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Golimumab 200 mg; Test type: Superiority or Other; p = 0.820, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p = 0.858, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change From Baseline in Domiciliary Morning Peak Expiratory Flow Rate (PEFR) at 6 Months; Randomized Subjects
Description: The endpoint is the change from baseline in domiciliary morning PEFR at Week 24. PEFR- Peak Expiratory Flow Rate (PEFR): A measure of the speed of exhalation. The data were collected in the eDiary which was issued to each participant at screening. PEFR was collected morning and evening each day of the study.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg | Combined: Group III & IV
Number analyzed (Participants) | 78 | 77 | 76 | 78 | 154
L/min | 4.730 (60.9136) | 8.102 (58.0602) | 3.488 (60.1336) | 2.475 (59.7923) | 2.975 (59.7668)
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group III & IV; The null hypothesis was that the endpoint for placebo is the same as that in the combined 100 mg and 200 mg golimumab; Test type: Superiority or Other; p = 0.833, ANOVA
Statistical Analysis 2: Comparison: Group I: Placebo vs Group IV: Golimumab 200 mg; Test type: Superiority or Other; p = 0.814, ANOVA
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p = 0.897, ANOVA
Statistical Analysis 4: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p = 0.726, ANOVA

ADVERSE EVENTS:
Groups:
- Group I: Placebo: Placebo subcutaneous (SC) injections every 4 wks from Wk 0 to Wk 52
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Group IV: Golimumab 200 mg
Serious Adverse Events (participants affected / at risk) | 16/78 | 24/75 | 24/78 | 22/78
Other Adverse Events (participants affected / at risk) | 75/78 | 68/75 | 75/78 | 75/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Placebo (N=78) | Group II: Golimumab 50 mg (N=75) | Group III: Golimumab 100 mg (N=78) | Group IV: Golimumab 200 mg (N=78)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 6 | 9
Diffuse panbronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 5 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 2
Sepsis (Infections and infestations) | 0 | 1 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Choriomeningitis lymphocytic (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Immune system disorders) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Hyperthermia (General disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Serum sickness (Immune system disorders) | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Borderline personality disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Placebo (N=78) | Group II: Golimumab 50 mg (N=75) | Group III: Golimumab 100 mg (N=78) | Group IV: Golimumab 200 mg (N=78)
Asthma (Respiratory, thoracic and mediastinal disorders) | 71 | 64 | 69 | 72
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 2
Sinusitis (Infections and infestations) | 9 | 19 | 17 | 10
Upper respiratory tract infection (Infections and infestations) | 16 | 7 | 14 | 12
Nasopharyngitis (Infections and infestations) | 10 | 9 | 8 | 12
Bronchitis (Infections and infestations) | 8 | 4 | 13 | 10
Rhinitis (Infections and infestations) | 5 | 3 | 5 | 6
Oral candidiasis (Infections and infestations) | 2 | 3 | 4 | 4
Influenza (Infections and infestations) | 4 | 1 | 5 | 4
Pneumonia (Infections and infestations) | 3 | 4 | 3 | 3
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 5
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 4
Acute sinusitis (Infections and infestations) | 7 | 2 | 1 | 1
Injection site erythema (General disorders) | 0 | 2 | 4 | 4
Pyrexia (General disorders) | 1 | 0 | 4 | 4
Chest pain (General disorders) | 5 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 3
Nausea (Gastrointestinal disorders) | 1 | 2 | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 4 | 3
Eczema (Skin and subcutaneous tissue disorders) | 5 | 2 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 1
Headache (Nervous system disorders) | 5 | 5 | 6 | 6
Migraine (Nervous system disorders) | 0 | 2 | 0 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 4 | 3

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <= 5% of patients. This information may vary from existing approved labeling and publications due to the requirement of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.